CLINICAL TRIAL: NCT00504348
Title: An Open-label Clinical Trial of the Combination Treatment of Tacrolimus and Corticosteroid in Polymyositis/Dermatomyositis Patients With Interstitial Pneumonitis, With Comparison Against Corticosteroid-treated Historical Controls
Brief Title: Investigation in Myositis-associated Pneumonitis of Prednisolone And Concomitant Tacrolimus
Acronym: IMPPACT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tokyo Medical and Dental University (Other)
Collaborators: Japan Medical Association (Industry); Astellas Pharma Inc (Industry)
Responsible Party: Principal Investigator, Kazuki Takada, MD, Professor, Institute of Education, Tokyo Medical and Dental University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IICT-FK506-01
Record Dates: First submitted 2007-07-19; First posted 2007-07-20 (Estimated); Results first posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Interstitial Pneumonitis; Polymyositis; Dermatomyositis
Keywords: Interstitial pneumonitis; Polymyositis; Dermatomyositis; Tacrolimus; Corticosteroids
MeSH Terms: conditions — Lung Diseases, Interstitial; Polymyositis; Dermatomyositis | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prospective investigation group (Experimental): Tacrolimus treatment is to be initiated at the starting dose of 0.075mg/kg/day, adjusted to maintain its whole blood trough levels between 5 and 10 ng/mL for 52 weeks. All patients are to receive glucocorticoids with the starting doses equivalent to between 0.6 and 1.0 mg/kg/day of prednisolone which are to be continued for the first 28 days after which be subsequently tapered according to a predefined guideline. Up to two courses of pulse intravenous glucocorticoid therapy are allowed during that period.
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Start at the standard starting dose of 0.075mg/kg/day divided into two doses, then adjust doses based on clinical response and tolerability, but maintain whole blood trough levels between 5 to 10 ng/mL and total daily doses equal to or below 0.3mg/kg.
  Other Names: Prograf

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of the combination treatment of tacrolimus and corticosteroid in polymyositis/dermatomyositis patients with interstitial pneumonitis with comparison against corticosteroid-treated historical controls.

DETAILED DESCRIPTION:
Interstitial pneumonia (IP) is a common complication of and has a significant impact on the prognosis of patients with polymyositis (PM) and dermatomyositis (DM). Reported prevalence of IP in PM/DM patients varies between 23 to 65% depending on criteria applied as well as on clinical settings of studied cohorts, and an earlier overview and a later study reported its high short-term mortality.

However, treatment for this grave complication has not yet been either established or even been prospectively investigated. Glucocorticoids, while long been considered as the first-line drugs, is effective in less than 50% of patients. Furthermore, the mortality of these glucocorticoids-resistant patients does not improve even if immunosuppressive drugs are later added.

Recently, we and others reported retrospective data which suggest that either an early addition of immunosuppressive drugs to glucocorticoids or the combined use of glucocorticoids and immunosuppressive drugs from the initial treatment may improve the survival of PM/DM patients. To save lives of PM/DM-IP patients, desperate treating physicians have started using this approach, strongly urging the conduct of prospective studies to investigate the superiority of this approach over glucocorticoids alone. At the same time, it was considered not ethically appropriate to conduct a prospective study with a concurrent controlled group receiving glucocorticoids alone given the presence of the PM/DM-IP subtype with rapidly progressive course and high short-term mortality if treated with glucocorticoids alone and the absence of useful demographic or bio-markers which could distinguish patients with this subtype early. Among immunosuppressive drugs used in the treatment of PM/DM-IP, tacrolimus has recently been suggested to be effective even for those patients who are resistant to cyclosporine or cyclosphosphamide.

To investigate whether the combined initial treatment of glucocorticoids and tacrolimus is superior to glucocorticoids alone in PM/DM-IP patients, we conducted a multicenter clinical trial to evaluate the efficacy and safety of a combination treatment of glucocorticoids and tacrolimus for 1 year in patients with newly developed active PM/DM-IP or its relapse by comparing against clinical outcome of historical control patients who were treated with glucocorticoid alone as an initial treatment.

ELIGIBILITY:
Inclusion Criteria:

Experimental treatment group

1. Diagnosis of definite or probable polymyositis or dermatomyositis by criteria of Bohan et al, or of clinically-amyopathic dermatomyositis by the definition proposed by Sontheimer et al
2. High-resolution CT findings consistent with interstitial pneumonitis, confirmed by a radiologist. If consolidation is the only abnormal findings, the patient must have pathologically documented evidence of interstitial pneumonitis of other histological type than cryptogenic organizing pneumonia/bronchiolitis obliterans organizing pneumonia (the patient could have more than one histological type including cryptogenic organizing pneumonia/bronchiolitis obliterans organizing pneumonia)
3. Meet two or more of the following criteria (must include 1) 1. Serum KL-6 above the upper normal limit 2. Presence of dyspnea on exertion (grade 2 on the Magnitude of Task component of the Mahler Modified Dyspnea Index 3. PaO2 of less than 80 mmHg while breathing ambient air at rest, not accompanied by abnormal increase of PaCO2 4. Vital capacity < 80% predicted, or diffusing capacity for carbon monoxide < 65% predicted 5. Meet at least one of the following condition over the 12-week period (84 days) prior to the initiation of the study drug

   * Decrease in either % forced vital capacity or % diffusing capacity for carbon monoxide of 10% or more
   * Worsening of interstitial pneumonitis findings by chest CT, confirmed by a radiologist
4. 16 to 74 years of age

Historical control group

1. Diagnosis of definite or probable polymyositis or dermatomyositis by criteria of Bohan et al, or of clinically-amyopathic dermatomyositis by the definition proposed by Sontheimer et al
2. High-resolution CT findings consistent with interstitial pneumonitis, confirmed by a radiologist. If consolidation is the only abnormal findings, the patient must have pathologically documented evidence of interstitial pneumonitis of other histological type than cryptogenic organizing pneumonia/bronchiolitis obliterans organizing pneumonia (the patient could have more than one histological type including cryptogenic organizing pneumonia/bronchiolitis obliterans organizing pneumonia)
3. Meet two or more of the following criteria (must include 1) 1. Serum KL-6 above the upper normal limit 2. Presence of dyspnea on exertion (grade 2 on the Magnitude of Task component of the Mahler Modified Dyspnea Index 3. PaO2 of less than 80 mmHg while breathing ambient air at rest, not accompanied by abnormal increase of PaCO2 4. Vital capacity < 80% predicted, or diffusing capacity for carbon monoxide < 65% predicted 5. Meet at least one of the following condition over the 12-week period (84 days) prior to the initiation of the study drug

   * Decrease in either % forced vital capacity or % diffusing capacity for carbon monoxide of 10% or more
   * Worsening of interstitial pneumonitis findings by chest CT, confirmed by a radiologist
4. Use of corticosteroids at doses equivalent to between 0.6 to 1.0mg/kg/day of prednisolone for 14 days or longer to treat interstitial pneumonitis on or after the day when the inclusion criteria (3) was met (up to two courses of pulse IV corticosteroid therapy within the first 28 days are allowed)
5. 16 to 74 years of age

Exclusion Criteria:

Experimental treatment group

1. Use of corticosteroids at doses equivalent to or higher than prednisolone 0.6mg/kg/day within 4 weeks (28 days) prior to the initiation of the study drug
2. Use of immunosuppressive agents other than corticosteroids within 12 weeks (84 days) prior to the initiation of the study drug
3. Could not exclude the following conditions on clinical ground: drug-induced pneumonitis, occupational lung disease, hypersensitivity pneumonitis, radiation-induced lung injury
4. Presence of end-stage interstitial pneumonitis as identified on the basis of a vital capacity < 45% predicted, diffusing capacity for carbon monoxide < 30% predicted, or lung CT with predominantly honeycombing appearance
5. Presence of pancreatitis
6. Presence of diabetes mellitus with the exception of glucocorticoid-induced one that is well-controlled (HbA1c < 6.5%)
7. Serum creatinine of 1.5 mg/dL or above
8. Presence of liver dysfunction (AST(GOT) or ALT (GPT) greater than 2.5 times the upper limit of normal) with the exception of the one that is considered to be due to myositis and is accompanied by the elevation of muscle enzymes above the upper limit of normal
9. Serum potassium above the upper limit of normal
10. Presence of ischemic heart disease, arrhythmia requiring treatment, congestive heart failure, or pulmonary hypertension requiring treatment
11. Presence or history of malignancy with the exception of those without relapse off treatment for 5 years or longer
12. Presence of serious active infection
13. Presence of active hepatitis B, hepatitis C, or HIV infection
14. History of severe drug hypersensitivity reaction
15. Patients who are pregnant or breast-feeding, or patients who intend to or whose spouses intend to conceive during the course of the study, including the follow-up period
16. Participation in another clinical trial or post-marketing clinical study within 26 weeks (182 days) prior to screening
17. Other medical condition which, in the investigator's judgment, may be associated with increased risk to the subject or may interfere with study assessments or outcomes

Historical control group

1. Use of immunosuppressive agents other than corticosteroids within 12 weeks (84 days) prior to or 2 weeks (14 days) after the corticosteroid treatment as defined by the inclusion criteria (4) is initiated
2. Could not exclude the following conditions on clinical ground: drug-induced pneumonitis, occupational lung disease, hypersensitivity pneumonitis, radiation-induced lung injury
3. Presence of end-stage interstitial pneumonitis as identified on the basis of a vital capacity < 45% predicted, diffusing capacity for carbon monoxide < 30% predicted, or lung CT with predominantly honeycombing appearance
4. Presence of pancreatitis
5. Presence of diabetes mellitus with the exception of glucocorticoid-induced one that is well-controlled (HbA1c < 6.5%)
6. Serum creatinine of 1.5 mg/dL or above
7. Presence of liver dysfunction (AST(GOT) or ALT (GPT) greater than 2.5 times the upper limit of normal) with the exception of the one that is considered to be due to myositis and is accompanied by the elevation of muscle enzymes above the upper limit of normal
8. Serum potassium above the upper limit of normal
9. Presence of ischemic heart disease, arrhythmia requiring treatment, congestive heart failure, or pulmonary hypertension requiring treatment
10. Presence or history of malignancy with the exception of those without relapse off treatment for 5 years or longer
11. Presence of serious active infection including active hepatitis B, hepatitis C, or HIV infection
12. Other medical condition which, in the investigator's judgment, may be associated with increased risk to the subject or may interfere with study assessments or outcomes

Ages: 16 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nobuyuki Miyasaka, MD, PhD, Principal Investigator — Tokyo Medical and Dental University
Locations (11):
- Japan (11):
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Tsukuba University Hospital, Tsukuba, Ibaraki
  - Osaka Minami Medical Center, Kawachi-Nagano, Osaka
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Tokyo Medical and Dental University Hospital, Bunkyo-ku, Tokyo
  - The University of Tokyo Hospital, Bunkyo-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - International Medical Center of Japan, Shinjuku-ku, Tokyo
  - Chiba University Hospital, Chiba
  - Nagasaki University Hospital of Medicine and Dentistry, Nagasaki
  - Tokushima University Hospital, Tokushima

REFERENCES:
- [Result] Takada K, Katada Y, Ito S, Hayashi T, Kishi J, Itoh K, Yamashita H, Hirakata M, Kawahata K, Kawakami A, Watanabe N, Atsumi T, Takasaki Y, Miyasaka N. Impact of adding tacrolimus to initial treatment of interstitial pneumonitis in polymyositis/dermatomyositis: a single-arm clinical trial. Rheumatology (Oxford). 2020 May 1;59(5):1084-1093. doi: 10.1093/rheumatology/kez394. PMID 31539061

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prospective Investigation Group
Started | 25
Completed | 17
Not Completed | 8
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 4
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Prospective Investigation Group
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival (OS) was calculated from the day on which the protocol treatment was started until death due to any cause. Participants still alive were censored at the date they were last known to be alive.
Time Frame: 52 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prospective Investigation Group
Number analyzed (Participants) | 25
percentage of participants | 88.0 [67.3 to 96.0]

2. Secondary Outcome: Progression-free Survival
Description: Patients were considered to have reached the progression if they died, or if they met all the following criteria; (1) ≥10% decline from baseline FVC or ≥15mmHg increase in baseline resting P(A-a)O2, (2) a worsening of interstitial pneumonitis findings by chest CT compared to the most recent study, confirmed by a radiologist, and (3) exclusion of pneumocystis pneumonia, cytomegalovirus pneumonia, and other pulmonary infection on clinical ground.
Time Frame: 52 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prospective Investigation Group
Number analyzed (Participants) | 25
percentage of participants | 76.4 [51.8 to 89.5]

ADVERSE EVENTS:
Time Frame: All adverse events observed between the first dose and 28 days after the last dose of tacrolimus.
Description: Testing for safety was performed at set intervals and consisted of vital signs and physical examinations, laboratory testing, and evaluation for adverse events and serious adverse events.
Arm/Group | Prospective Investigation Group
All-Cause Mortality (participants affected / at risk) | 4/25
Serious Adverse Events (participants affected / at risk) | 11/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prospective Investigation Group (N=25)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 6
zoster (Skin and subcutaneous tissue disorders) | 1
Nocardiosis (Infections and infestations) | 1
Cytomegalovirus pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumocystis jiroveci pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Cataract (Eye disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Liver cirrhosis (Hepatobiliary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prospective Investigation Group (N=25)
Nasopharyngitis (Infections and infestations) | 6 (8)
Zoster (Infections and infestations) | 4 (5)
Bronchitis (Infections and infestations) | 2 (2)
Cystitis (Infections and infestations) | 2 (2)
Gastroenteritis (Infections and infestations) | 2 (2)
Onychomycosis (Infections and infestations) | 2 (2)
Oral candidiasis (Infections and infestations) | 2 (2)
Pharyngeal candidiasis (Infections and infestations) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Cushingoid appearance (Endocrine disorders) | 5 (5)
Diabetes mellitus (Endocrine disorders) | 7 (8)
Dyslipidemia (Endocrine disorders) | 7 (7)
Glucose intolerance (Endocrine disorders) | 6 (6)
Hyperkalemia (Endocrine disorders) | 4 (4)
Hypoglycemia (Endocrine disorders) | 3 (3)
Dehydration (Endocrine disorders) | 2 (2)
Hypomagnesemia (Endocrine disorders) | 2 (2)
Hypophosphatemia (Endocrine disorders) | 2 (2)
Hyperlipidemia (Endocrine disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 5 (6)
Tremor (Nervous system disorders) | 7 (7)
Hypesthesia (Nervous system disorders) | 3 (5)
Dizziness (Nervous system disorders) | 2 (2)
Cataract (Eye disorders) | 2 (2)
Conjunctival hemorrhage (Eye disorders) | 2 (2)
Conjunctivitis (Eye disorders) | 2 (2)
Ventricular extrasystole (Cardiac disorders) | 3 (3)
Hypertension (Vascular disorders) | 6 (8)
Hypotension (Vascular disorders) | 2 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 9 (9)
Diarrhea (Gastrointestinal disorders) | 6 (7)
Stomatitis (Gastrointestinal disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Upper abdominal pain (Gastrointestinal disorders) | 2 (2)
Cheilitis (Gastrointestinal disorders) | 2 (2)
Colon polyp (Gastrointestinal disorders) | 2 (2)
Erosive gastritis (Gastrointestinal disorders) | 2 (2)
Fatty liver (Hepatobiliary disorders) | 2 (2)
Liver disorder (Hepatobiliary disorders) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 4 (4)
Subcutaneous hemorrhage (Skin and subcutaneous tissue disorders) | 4 (5)
Skin rash (Skin and subcutaneous tissue disorders) | 3 (3)
Skin abrasion (Skin and subcutaneous tissue disorders) | 3 (3)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2)
Asteatotic eczema (Skin and subcutaneous tissue disorders) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Onycholysis (Skin and subcutaneous tissue disorders) | 2 (2)
Myopathy (Musculoskeletal and connective tissue disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Renal dysfunction (Renal and urinary disorders) | 3 (3)
Peripheral edema (General disorders) | 4 (4)
Feeling unwell (General disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Conclusion is not based on meaningful statistical comparison, will not apply to asymptomatic or subclinical IP, or to the exacerbation of IP, or will not separately provide the efficacy of the treatment in the anti-MDA-5 positive subgroup.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No